CLINICAL TRIAL: NCT03808116
Title: Evaluation of the SmartBx System for Breast Biopsy Download While Keeping the Orientation, Unfolding and Unity of the Sample
Brief Title: Evaluation of the SmartBx System for Breast Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UC Care, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EMC-0124-18
Record Dates: First submitted 2019-01-09; First posted 2019-01-17 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer
Keywords: breast biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SmartBx biopsy collection (Experimental): * Biopsy cores will be collected from the breast during US guided biopsy procedure.
  * The number of cores taken will be decided per the physician discretion according to the clinical demand.
  * Additional two biopsy core will be taken the SmartBx cassette
  Interventions: Device: SmartBx

INTERVENTIONS:
Device: SmartBx — he SmartBx device is intended for the retention of a biopsy specimen and for preservation of the specimen's in-needle location and orientation.
  The SmartBx is used as an aiding tool in biopsy procedures. When operated in conjunction with the standard equipment in a prostate biopsy procedure, the SmartBx may be used for the following:
  * To preserve sample unity, including core fragments in their original location along the needle notch.
  * Avoid sample damaging during sample removal from the needle and the following pathology process.

SUMMARY:
Performance evaluation of a novel, semi-automated device and method for needle core biopsy download compared to standard methods in terms of:

3. Biopsy core length obtained (i.e. collecting all tissue fragments) 4. Biopsy core yield (i.e. percent of tissue loss during the pathologic processing)

DETAILED DESCRIPTION:
Examination procedure:

* Biopsy cores will be collected from the breast during US guided biopsy procedure.
* The number of cores taken will be decided per the physician discretion according to the clinical demand.
* Additional two biopsy core will be taken the SmartBx cassette. Since the SmartBx cassette holds two biopsies together, two consecutive cores will be collected using the SmartBx.
* samples will be photographed for measurements in 2 steps during the process:

  1. On the needle notch [A].
  2. On the glass slide [B].
* Standard tissue fixation, processing of the samples in paraffin will be performed unchanged per the pathology laboratory protocols.
* Embedding of the biopsy cores taken with the SmartBx will be embedded using the SmartBx mold and tamper.
* Standard staining and histology analysis will be preformed to the sectioned samples, unchanged per the pathology protocols.

  • Analysis will be preformed to the histological results, and a comparison between the standard procedures samples to the SmartBx samples will be performed in terms of -
* Biopsy core length obtained (i.e. collecting all tissue fragments)
* Biopsy core yield (i.e. percent of tissue loss during the pathologic processing)

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Planned for breast biopsy procedure.
* Signed informed consent.

Exclusion Criteria:

o Patient's unwilling to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
biopsy core length | 1 month
  biopsy core length will be measured on the glass slide
biopsy core yield | 1 month
  biopsy core length will be measured on the needle and on the glass slide and for each core the length on the slide will be computed in reference to the length on the needle

CONTACTS AND LOCATIONS:
Locations (1):
- Haemek medical center, Afula, North Region, Israel